CLINICAL TRIAL: NCT00727675
Title: Chronic Pain and Opioid Dependence Assessment and Treatment
Acronym: CPODAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0703002496; 1K23DA024050-01A1 (NIH)
Record Dates: First submitted 2008-07-31; First posted 2008-08-04 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Chronic Pain; Opioid Dependency
Keywords: chronic pain; opioid dependence; Cognitive Behavioral Therapy (CBT)
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Integrated Cognitive Behavioral Therapy for pain reduction and opioid dependence.
  Interventions: Behavioral: Integrated Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Integrated Cognitive Behavioral Therapy — CBT is provided by skilled psychologists in weekly sessions for 12 weeks and focuses on reducing illicit drug use and increasing pain management.

SUMMARY:
This study involves the development of an integrated psychotherapy that addresses both chronic pain and opioid dependence(POD).

DETAILED DESCRIPTION:
To conduct a pre-pilot study with 20 POD patients to a) evaluate the acceptability and potential efficacy of specific sessions (i.e., reduced illicit opioid use as assessed by urine toxicology and self-report findings, and decreased pain as evidenced by attenuated pain intensity and pain interference on self-report measures from baseline throughout treatment) for inclusion in integrated Cognitive Behavioral Therapy (CBT) for POD and the sequence of sessions, b) assess patients' satisfaction with integrated CBT as evidenced by qualitative feedback from individual exit interviews, and c) develop and modify initial therapist training and process rating measures. Products will include a) a manual for integrated CBT for POD to be used in opioid treatment programs and primary care settings with POD patients, b) therapist training materials, and c) process rating instruments.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* currently in Methadone Maintenance Treatment (MMT) at the APT Foundation in New Haven, CT
* opioid dependence
* experience moderate to severe chronic pain

Exclusion Criteria:

* current suicide or homicide risk
* are unable to complete the informed consent or surveys because of psychiatric impairment
* have cognitive impairment
* are unable to read or understand English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-08; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Reduced illicit opioid use and pain | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Declan T. Barry, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Barry DT, Cutter CJ, Beitel M, Kerns RD, Liong C, Schottenfeld RS. Psychiatric Disorders Among Patients Seeking Treatment for Co-Occurring Chronic Pain and Opioid Use Disorder. J Clin Psychiatry. 2016 Oct;77(10):1413-1419. doi: 10.4088/JCP.15m09963. PMID 27574837